CLINICAL TRIAL: NCT02355171
Title: A Large-scale Longitudinal Oncology Registry
Brief Title: Personalize My Treatment (PMT) Registry
Acronym: PMT
Status: Suspended | Type: Observational
Why Stopped: Biobank - no investigation involved
Sponsor: Exactis Innovation (Other)
Responsible Party: Sponsor
Other Study IDs: PMT
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tissue (from surgical resection or biopsy) and blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The 'Personalize My treatment' (PMT) platform is a novel form of biobanking in which cancer patients willingly consent to provide residual, clinical samples (surplus after diagnostic testing) of their tumors for cancer research, to give access to their medical record for data collection and then followed prospectively throughout the trajectory of their illness. They further willingly consent to be recontacted for being informed of other research projects, including clinical trials.

ELIGIBILITY:
Age of majority in the province of recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with all solid tumor types.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-11; Primary Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
The primary objective of PMT is to create a collection of cancer patient biospecimens and annotated data that will be used for clinical trial matching and to advance cancer research. | Longitudinal

CONTACTS AND LOCATIONS:
Locations (14):
- Canada (14):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Centre Hospitalier Universitaire Dr-Georges-L.-Dumont, Moncton, New Brunswick
  - The Moncton Hospital, Moncton, New Brunswick
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Science Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Odette Cancer Centre - Sunnybrook Hospital, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - MUHC McGill University Health Center, Montreal, Quebec
  - Centre hospitalier universitaire de Québec - Université Laval, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - CIUSSS de la Mauricie-et-du-Centre-du-Québec - Centre Hospital Régional, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: Yes
The BDAC (Biospecimen and Data Access Committee) authorizes access requests from researchers to the PMT Platform's biospecimens and data. It meets as needed to review requests in accordance with the PMT Biospecimen and Data Access Policy. Requests will be evaluated based on scientific merit, availability of sample and alignment with the mission of the PMT Platform and Exactis. BDAC is responsible for verifying that the proposed project has received appropriate ethics approval and proof of such approval has been provided.

REFERENCES:
- See also: exactis.ca — https://www.exactis.ca